CLINICAL TRIAL: NCT00441038
Title: Controlled Randomized Clinical Trial on the Effect on Low Back Pain Related Disability of Different Health Education Programs for Retired Persons
Brief Title: A Trial on the Effect on Low Back Pain Related Disability of Different Health Education Programs for Retired Persons
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study showed recruitment rates were lower than expected,and number of losses to follow-up, much higher.
Sponsor: Kovacs Foundation (Other)
Collaborators: Conseill Insular de Ibiza y Formentera (Unknown); Mallorca Institute of Social Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FK-R-13
Record Dates: First submitted 2007-02-23; First posted 2007-02-28 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; disability; health education
MeSH Terms: conditions — Low Back Pain; Health Education | interventions — Blood Circulation; Health Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Education on postural hygiene and handout of The Back Guide
  Interventions: Behavioral: The Back Guide; Behavioral: The Back Book; Behavioral: Cardiovascular and general health
- 2 (Active Comparator): Education on active management and handout of The Back Book
  Interventions: Behavioral: The Back Book; Behavioral: Cardiovascular and general health
- 3 (Active Comparator): Education on cardiovascular and general health
  Interventions: Behavioral: Cardiovascular and general health

INTERVENTIONS:
Behavioral: The Back Guide — Education on postural hygiene and handout of The Back Guide
  Arms: 1
Behavioral: The Back Book — Education on active management and Handout of The Back Book
  Arms: 1; 2
Behavioral: Cardiovascular and general health — Education on cardiovascular and general health

SUMMARY:
The primary purpose of this study is to compare, in retired persons living in the Balearic Islands, the effectiveness on low back pain related disability of three educational programs. All consist of a group talk and the handout of a booklet, each one different in its content.

ELIGIBILITY:
Inclusion Criteria:

* To attend regular talks for retirees, and accept to attend one health talk, whether or not subject has nonspecific low back pain; to accept participation in the study.

Exclusion Criteria:

* Inability to fill out questionnaires (due to blindness, functional illiteracy, or dementia);
* Having a diagnosis of rheumatologic inflammatory disease, fibromyalgia, or cancer in last 5 years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain, measured at baseline, 30, and 180 days | 6 months
Disability, measured at baseline, 30, and 180 days | 6 months

SECONDARY OUTCOMES:
Fear avoidance beliefs, measured at baseline, 30, and 180 days | 6 months
Quality of life, measured at baseline, 30, and 180 days | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M. Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; Juan Noguera, MD, Principal Investigator — Instituto de Asuntos Sociales y Deportes de Mallorca, Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Cherkin DC, Eisenberg D, Sherman KJ, Barlow W, Kaptchuk TJ, Street J, Deyo RA. Randomized trial comparing traditional Chinese medical acupuncture, therapeutic massage, and self-care education for chronic low back pain. Arch Intern Med. 2001 Apr 23;161(8):1081-8. doi: 10.1001/archinte.161.8.1081. PMID 11322842
- [Background] Indahl A, Haldorsen EH, Holm S, Reikeras O, Ursin H. Five-year follow-up study of a controlled clinical trial using light mobilization and an informative approach to low back pain. Spine (Phila Pa 1976). 1998 Dec 1;23(23):2625-30. doi: 10.1097/00007632-199812010-00018. PMID 9854762
- See also: Spanish Back Pain Research Network site that describes objectives and projects of its members — http://www.reide.org